CLINICAL TRIAL: NCT04704336
Title: Integration of Hypertension Management Into HIV Care in Nigeria: A Task Strengthening Strategy
Brief Title: Integration of Hypertension Management Into HIV Care in Nigeria
Acronym: TASSH NIMR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-00009; R01HL147811-01A1 (NIH)
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Human Immunodeficiency Virus; Hypertension
Keywords: Hypertension; Implementation science research; Integrated models; Practice Facilitation; People living with HIV; Human Immunodeficiency Virus; Cluster trial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypertension | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-directed without Practice Facilitation (PF) (No Intervention): Participants will be identified from HIV clinics during routine visits and provided standard of care.
- With Practice Facilitation (PF) (Experimental): Participants will be identified from HIV clinics during routine visits and will receive the task-shifting strategy for HTN control (TASSH) protocol.
  Interventions: Behavioral: Task-shifting strategy for HTN control (TASSH) protocol

INTERVENTIONS:
Behavioral: Task-shifting strategy for HTN control (TASSH) protocol — The TASSH protocol include the following 4 steps: 1). Identify HIV patients with uncontrolled HTN: trained HIV nurses will take patients' medical history (whether or not they have a diagnosis of diabetes, heart attack, stroke, heart failure, smoking). 2) Next, they will measure the patients' weight, height, waist circumference and BP with a valid automated device following standard procedures and then conduct lab tests with point-of-care testing on blood glucose, lipids and urine dip stick. 3) Initiate lifestyle counseling and medication treatment every 1-3 months: The nurses will next counsel eligible patients on lifestyle behaviors for 20 to 30 minutes (increased intake of fruits and vegetables, moderate physical activity and reduce salt intake). 4). Refer patients with complicated HTN to physicians for further care
  Arms: With Practice Facilitation (PF)

SUMMARY:
This study evaluates a tailored-practice facilitation (PF) strategy for integrating a task strengthening strategy for hypertension control (TASSH) for the care of patients living with HIV (PWH) within primary health centers (PHCs) in Lagos, Nigeria.

DETAILED DESCRIPTION:
Although access to antiretroviral therapy has led to increased survival among people living with HIV (PWH) in Africa, this population now has higher cardiovascular disease (CVD) - mortality than the general population largely due to an increased burden of hypertension. In Nigeria, the acute shortage of physicians limits the capacity to control hypertension among PWH at the primary care level where the majority receive treatment. This study proposes the use of practice facilitation (PF) - which will provide external expertise on practice redesign and a tailored approach to delivery of the evidence-based task strengthening strategy - to integrate hypertension into the HIV care model. Using a clinical-effectiveness implementation design, we will evaluate the effect of a PF strategy for integrating an evidence-based intervention for hypertension (HTN) control into HIV care among 960 patients with uncontrolled HTN in 30 primary health centers (PHCs) in Nigeria. Study is in 3 phases: 1) a pre-implementation phase that will develop a tailored PF intervention for integrating TASSH into HIV clinics; 2) an implementation phase that will compare the clinical effectiveness of PF vs. a self-directed condition (receipt of information on TASSH without PF) on BP reduction; and 3) a post- implementation phase to evaluate the effect of PF vs. self-directed condition on the adoption and sustainability of TASSH. The PF intervention comprises: (a) an advisory board to provide leadership support for implementing TASSH in HIV clinics; (b) training of the HIV nurses on TASSH protocol; and (c) training of practice facilitators, who will serve as coaches, provide support, and performance feedback to the HIV nurses

ELIGIBILITY:
Inclusion Criteria:

* Be an adult aged 18 years and older.
* Attends one of the 30 HIV clinics.
* Have a diagnosis of HTN with uncontrolled blood pressure, i.e. BP is 140-179/90-100 mm Hg.
* Ability to provide consent.

Exclusion Criteria:

* BP>180/110 mm Hg;
* history of chronic kidney disease, heart disease, diabetes or stroke, pregnancy
* Inability to provide informed consent.
* Refusal to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Olugbenga Ogedegbe, MD, Principal Investigator — NYU Langone Health
Locations (2):
- Saint Louis University (SLU), St Louis, Missouri, United States
- Nigerian Institute of Medical Research (NIMR), Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.To achieve aims in the approved proposal. For individual participant data meta-analysis. Requests should be directed to Olugbenga.Ogedegbe@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Iwelunmor J, Ezechi O, Obiezu-Umeh C, Oladele D, Nwaozuru U, Aifah A, Gyamfi J, Gbajabiamila T, Musa AZ, Onakomaiya D, Rakhra A, Jiyuan H, Odubela O, Idigbe I, Engelhart A, Tayo BO, Ogedegbe G. Factors influencing the integration of evidence-based task-strengthening strategies for hypertension control within HIV clinics in Nigeria. Implement Sci Commun. 2022 Apr 15;3(1):43. doi: 10.1186/s43058-022-00289-z. PMID 35428342
- [Derived] Aifah AA, Odubela O, Rakhra A, Onakomaiya D, Hu J, Nwaozuru U, Oladele DA, Odusola AO, Idigbe I, Musa AZ, Akere A, Tayo B, Ogedegbe G, Iwelunmor J, Ezechi O. Integration of a task strengthening strategy for hypertension management into HIV care in Nigeria: a cluster randomized controlled trial study protocol. Implement Sci. 2021 Nov 16;16(1):96. doi: 10.1186/s13012-021-01167-3. PMID 34789277

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Primary Health Centers (PHCs)
Period: Overall Study
Arm/Group | Self-directed Without Practice Facilitation (PF) | With Practice Facilitation (PF)
Started | 353; 15 Primary Health Centers (PHCs) | 477; 15 Primary Health Centers (PHCs)
Completed | 318; 15 Primary Health Centers (PHCs) | 435; 15 Primary Health Centers (PHCs)
Not Completed | 35; 0 Primary Health Centers (PHCs) | 42; 0 Primary Health Centers (PHCs)
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 33 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-directed Without Practice Facilitation (PF) | With Practice Facilitation (PF) | Total
Number analyzed (Participants) | 353 | 477 | 830
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (9.4) | 49.1 (9.6) | 49.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 289 | 527
  Male | 115 | 188 | 303
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 353 | 477 | 830
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 353 | 477 | 830
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Nigeria | 353 | 477 | 830

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: The primary outcome is change in systolic blood pressure (SBP) from baseline to 12 months. Following the research investigators' existing TASSH protocol, the SBP reduction in patients will assessed as mean change in systolic BP from baseline to 12 months. Blood pressure will be taken with valid automated BP device from the existing TASSH protocol.
Time Frame: Baseline, Month 12
Measure: Mean (95% Confidence Interval); unit: Change in SBP (mmHg)
Arm/Group | Self-directed Without Practice Facilitation (PF) | With Practice Facilitation (PF)
Number analyzed (Participants) | 353 | 477
Change in SBP (mmHg) | -12.8 [-14.9 to -10.7] | -15.1 [-16.5 to -13.7]

2. Secondary Outcome: Rate of Adoption of TASSH Across PHCs at 12 Months
Description: Rate of adoption of TASSH is defined as the proportion of patients who were diagnosed with HTN by the HIV nurses; received lifestyle counseling and antihypertensive treatment from HIV nurses. For this purpose, adoption will be assessed as a composite of the following measures: 1) the number of hypertensive patients diagnosed by the nurses using the WHO CVD risk assessment; 2) proportion of patients with HTN who received lifestyle counseling from the nurses; and 3) proportion of patients for whom the HIV nurses initiated treatment with antihypertensive medications. In order to assess this measure, the nurses will complete a questionnaire inquiring about the number of patients with uncontrolled HTN who received medication treatment and lifestyle counseling.
Time Frame: Month 12
Reporting Status: Not Posted

3. Secondary Outcome: Sustainability of TASSH Across PHCs at 24 Months
Description: Sustainability of TASSH is defined as the maintenance of TASSH uptake at the HIV clinics at 24 months (one year after the end of the intervention). Sustainability will be assessed with a composite quantitative measure similar to adoption and qualitatively, based on interviews with nurses and clinic leadership at 24 months. For this purpose, two research coordinators will conduct the interviews with two nurses and one key leadership personnel at each primary health center (PHCs).
Time Frame: Month 24
Reporting Status: Not Posted

4. Secondary Outcome: Implementation Climate Across PHCs at 12 Months
Description: Implementation Climate will be assessed with the Implementation Climate Scale. It measures shared perceptions of policies, practices, procedures, and behaviors that are expected, supported, and rewarded to facilitate effective evidence-based practice (EBP) implementation. It is an 18-item questionnaire that comprises six subscales. Each item is rated on a 5-point Likert scale from 0-4; each subscale score is calculated as the mean score of the associated items; the total score is the average of the six subscale scores and ranges from 0-4. Higher scores indicate a climate that is highly supportive of implementing EBPs.
Time Frame: Month 12
Reporting Status: Not Posted

5. Secondary Outcome: Implementation Climate Across PHCs at 24 Months
Description: as for outcome 4
Time Frame: Month 24
Reporting Status: Not Posted

6. Secondary Outcome: Implementation Leadership Across PHCs at 12 Months
Description: Implementation Leadership will be assessed with the Implementation Leadership Scale (ILS). It is a 12-item measure with four subscales: Proactive Leadership (α=.95), Knowledgeable Leadership (α=.96), Supportive Leadership (α=.95), and perseverant leadership (α=.96) and a total score (α=.98). Each item is rated on an item-specific Likert scale. Each subscale score is calculated as the mean score of the associated items; the total score is the average of the four subscale scores and ranges from 0-4. Higher scores indicate greater implementation leadership.
Time Frame: Month 12
Reporting Status: Not Posted

7. Secondary Outcome: Implementation Leadership Across PHCs at 24 Months
Description: as for outcome 6
Time Frame: Month 24
Reporting Status: Not Posted

8. Secondary Outcome: Change in Proficiency Across PHCs at 12 Months
Description: Proficiency will be assessed using the Organizational Culture domain of the Organizational Social Context Scale, a 15-item Proficiency subscale used to evaluate the practice capacity proficiency level of the primary health centers (PHCs). Proficient Organizational Cultures are those characterized by shared norms and expectations that the nurses are skilled service providers, and have current knowledge of the TASSH protocol. Items are completed using a 5-point rating scale ranging from 1 (never) to 5 (always) with measures such as responsiveness (e.g., 'members of my organizational unit are expected to be responsive to the needs of each patient') and competence (e.g., 'members of my organizational unit are expected to have up-to-date knowledge'). The total score is the sum of responses and ranges from 15-75; higher scores indicate more proficient organizational cultures. Alpha reliability for the proficient culture scale is .89.
Time Frame: Month 12
Reporting Status: Not Posted

9. Secondary Outcome: Change in Proficiency Across PHCs at 24 Months
Description: as for outcome 8
Time Frame: Month 24
Reporting Status: Not Posted

10. Secondary Outcome: Change in Organizational Readiness to Change - Evidence Across PHCs at 12 Months
Description: Organizational Readiness to Change - Evidence is assessed with the 12-item Evidence Scale, which evaluates the strength of the evidence for the proposed change/innovation. It will be used to evaluate intervention process measures focused on CFIR's Evidence Strength & Quality and Relative Advantage construct. Each item measures the extent to which a respondent agrees or disagrees with the item statement on a 5-point Likert- type scale (1 = strongly disagree; 5 = strongly agree) and the Cronbach α=0.74. The total score is the sum of responses and ranges from 12 to 60; higher scores indicate greater strength of the evidence for the proposed change/innovation.
Time Frame: Month 12
Reporting Status: Not Posted

11. Secondary Outcome: Change in Organizational Readiness to Change - Evidence Across PHCs at 24 Months
Description: as for outcome 10
Time Frame: Month 24
Reporting Status: Not Posted

12. Secondary Outcome: Change in External Change Agent Support Across PHCs at 12 Months
Description: External change agent support is assessed using a 3-item tool that evaluates support provided by external facilitators, the expectations about performance and improvement, and the ways to achieve the goal of the project. Items are scored on a 5-point Likert scale from 1-5 and the Cronbach α=0.77. The total score is the sum of responses and ranges from 3-15; higher scores indicate greater external change agent support.
Time Frame: Month 12
Reporting Status: Not Posted

13. Secondary Outcome: Change in External Change Agent Support Across PHCs at 24 Months
Description: as for outcome 12
Time Frame: Month 24
Reporting Status: Not Posted

14. Secondary Outcome: Change in Organizational Readiness to Change - Facilitation Across PHCs at 12 Months
Description: Organizational Readiness to Change - Facilitation is measured using the Facilitation Scale (8-items) evaluates organizational capacity to facilitate change will be used to evaluate implementation process measures focused on CFIR Engaging construct. Each item measures the extent to which a respondent agrees or disagrees with the item statement on a 5-point Likert-type scale (1 = strongly disagree; 5 = strongly agree). It has Cronbach α=0.95. The total score is the sum of responses and ranges from 8-40; higher scores indicate greater organizational capacity to facilitate change.
Time Frame: Month 12
Reporting Status: Not Posted

15. Secondary Outcome: Change in Organizational Readiness to Change - Facilitation Across PHCs at 24 Months
Description: as for outcome 14
Time Frame: Month 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Follow-up until end of Month 24.
Description: Non-systematic.
Arm/Group | Self-directed Without Practice Facilitation (PF) | With Practice Facilitation (PF)
All-Cause Mortality (participants affected / at risk) | 6/353 | 4/477
Serious Adverse Events (participants affected / at risk) | 4/353 | 8/477
Other Adverse Events (participants affected / at risk) | 2/353 | 0/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Self-directed Without Practice Facilitation (PF) (N=353) | With Practice Facilitation (PF) (N=477)
Cerebrovascular accident (CVA) (Nervous system disorders) | 1 | 3
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 3 | 0
Bell's Palsy (Nervous system disorders) | 0 | 1
Kidney Problem (Renal and urinary disorders) | 0 | 1
Chronic Left Leg Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Self-directed Without Practice Facilitation (PF) (N=353) | With Practice Facilitation (PF) (N=477)
Diarrheal Disease (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04704336/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT04704336/ICF_000.pdf